CLINICAL TRIAL: NCT02225054
Title: The Analgesic Effect of Dexmedetomidine as an Adjunct to Local Anesthetics in Ultrasound-guided Interscalene Approach to Brachial Plexus Block for Shoulder Surgery: A Randomized Controlled Trial
Brief Title: The Effect of Dexmedetomidine on Brachial Plexus Block for Shoulder Surgery
Acronym: DEX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DEX-2013
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Nerve Pain; Shoulder Pain
Keywords: duration of analgesia
MeSH Terms: conditions — Neuralgia; Shoulder Pain | interventions — Dexmedetomidine; Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ropivacaine,Normal Saline,Saline Bolus (Placebo Comparator): Ropivacaine 15 mL 0.5% Normal Saline mL 0.9% Saline Bolus
  Interventions: Drug: Ropivacaine; Drug: Normal Saline
- Ropivacaine,Dexmedetomidine,Saline Bolus (Experimental): Ropivacaine15 mL 0.5% Dexmedetomidine0.5 u/kg Saline Bolus
  Interventions: Drug: Dexmedetomidine; Drug: Ropivacaine; Drug: Normal Saline
- Ropivacaine,Saline,Dexmedetomidine (Active Comparator): Ropivacaine 15 mL 0.5% Normal Saline 1 mL 0.9% Dexmedetomidine single IV bolus 0.5 u/kg over 30 minutes
  Interventions: Drug: Dexmedetomidine; Drug: Ropivacaine; Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine — 0.5 u/kg Dexmedetomidine diluted in saline to 1 mL (single interscalene injection) Dexmedetomidine 0.5 u/kg as a single IV bolus over 30 minutes following GA induction
  Other Names: Precedex
  Arms: Ropivacaine,Dexmedetomidine,Saline Bolus; Ropivacaine,Saline,Dexmedetomidine
Drug: Ropivacaine — 15 ml 0.5%
  Other Names: Naropin
Drug: Normal Saline — 1 mL 0.9%

SUMMARY:
The purpose of this study is to determine whether a small dose of Dexmedetomidine, when given either intravenously or as part of the interscalene nerve block solution, prolongs pain relief following shoulder surgery compared to local anesthetic solution alone.

DETAILED DESCRIPTION:
Unilateral shoulder surgical procedures, including acromioplasty, rotator cuff repair and Bankart procedure generally allow the patient to go home the same day. However, post-surgical pain is often severe and it is common to encounter a delay in discharge from the hospital due to difficulty in pain control.

Single shot interscalene block is used in ambulatory shoulder surgery for its advantages that included a significant reduction in acute pain and analgesic requirements, prolonged time to first analgesic request, decreased incidence of nausea, as well as earlier hospital discharge. Previous studies have attempted to prolong the duration of the analgesia of interscalene block by administering additional drugs to the local anesthetics but these studies have had varying degrees of success. Dexmedetomidine has recently been considered as a potentially useful drug in prolonging nerve block analgesia. Various modes of administration of Dexmedetomidine have demonstrated a consistent effect on the duration of analgesia. So far, the systemic infusion of Dex has been shown to prolong both neuraxial and peripheral nerve blocks. When combined with local anesthetics in intravenous regional anesthesia 9IVRA), Dex enhanced the duration of analgesia. Furthermore, data from animal studies strongly support the use of Dex as a safe potent adjunct to local anesthetics capable of prolonging the duration of analgesia of peripheral nerve blocks.

The use of Dexmedetomidine as an adjunct in interscalene block has not been studied yet. This trial will study the effects of adding Dexmedetomidine as an adjunct to local anesthetics in interscalene brachial plexus block.

ELIGIBILITY:
Inclusion Criteria:

* unilateral surgical shoulder procedures under general anesthetic
* English speaking patients
* ASA I-III patients
* BMI <38 kg/m2

Exclusion Criteria:

* proximal clavicular surgery
* preexisting neurological deficits or peripheral neuropathy
* known coronary heart disease, congestive heart failure, cardiomyopathies, or arrhythmias
* known cerebrovascular disease
* baseline heart rate <60 beats per minute or baseline systolic blood pressure <100 mm Hg
* medications that reduce heart rate (as beta-blockers, calcium blockers) known liver dysfunction or existing diseases known to cause hepatic or renal impairment
* severe bronchopulmonary disease
* local infection
* contra-indication to regional anesthesia (bleeding, coagulopathy)
* chronic pain disorders
* current use of over 30mg oxycodone or equivalent per day
* contraindication to a component of multimodal analgesia
* allergy to local anesthetics or dexmedetomidine
* history of significant psychiatric conditions that may affect patient assessment
* pregnancy
* inability to provide consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Duration of interscalene nerve block. | Duration of time is from the end of local anesthetic injection (interscalene block) to the onset of pain at the surgical site.
Opioid consumption | Cumulative opioid consumption at 24 hours postoperatively

SECONDARY OUTCOMES:
Opioid Consumption | Total use of opioids from the period of intra-operative to 2 weeks post-operative
  The total amount of opioid use starting from during surgery to 14 days following surgery. Opioid side effects, patient satisfaction with pain control and the time to discharge from hospital will all be assessed Any evidence of nerve block complications at 3 months, post-block administration , will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Richard M. Brull, MD, FRCPC, Principal Investigator — University of Toronto, Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada